CLINICAL TRIAL: NCT04798417
Title: Nutrition to Relieve IBS Constipation
Acronym: NUTRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: Ministery of Economic affairs (Unknown); Nexira (Industry); Wecare (Other); Roquette Freres (Industry); Ingredion Incorporated (Industry); Ingredia S.A. (Industry); Naturex (Other); Winclove Probiotics B.V. (Industry); Bioiberica (Industry); Darling Ingredients (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL76449.041.21
Record Dates: First submitted 2021-03-04; First posted 2021-03-15 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Irritable Bowel Syndrome; Constipation
Keywords: Prebiotic; Probiotic
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic supplement
- Prebiotic (Experimental)
  Interventions: Dietary Supplement: Prebiotic supplement
- Maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — Use of a probiotic sachet
  Arms: Probiotic
Dietary Supplement: Prebiotic supplement — Prebiotic sachets
  Arms: Prebiotic
Dietary Supplement: Maltodextrin — Placebo comparator
  Arms: Maltodextrin

SUMMARY:
Rationale: Irritable Bowel Syndrome (IBS) is a disease that affects a large number of people. To date, no adequate treatment is available. This is partially due to the heterogeneity of the patients and the complicated pathology in which not all mechanisms are understood. Based on results of in vitro screening within the IBSQUtrition project, we selected promising dietary supplements for validation of their potential beneficial effects on stool pattern in IBS-Constipation (IBS-C) patients.

Objective: The primary objective is to determine the effects of a 4-week intervention with either a prebiotic supplement or a probiotic supplement on stool pattern (including stool frequency, consistency, and volume) in IBS-C patients. The secondary objective is to determine the effects if this intervention on GI complaints and quality of life in IBS-C patients.

Study design: A double-blind, randomized, placebo-controlled trial will be conducted with three parallel intervention arms Study population: 180 adult (18-70 yrs) IBS patients with a constipation-predominant subtype Intervention: A 4 week run-in period will be followed by a 4-week intervention period with three parallel arms: 1) prebiotic supplement, 2) probiotic supplement, and 3) Placebo supplement, during which the study participants consume the respective supplement twice per day.

Main study parameters/endpoints: The primary study parameter is stool pattern: stool frequency, stool consistency; and stool volume. The secondary study parameters are gastrointestinal complaints, Quality of Life, and HADS.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Study participants have to invest about 14.5 hours of their time in this study mainly to complete several questionnaires (short daily questionnaire, longer questionnaires at three occasions), which is conveniently all possible from home. They have to comply to consume a supplement twice daily for four weeks. At two time points they have to collect their stool for five consecutive days. There are limited risks for the study participants.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients that meet the Rome IV criteria + additional criteria specific for the constipation-predominant subtype, based on the most frequent self-reported stool types using the Bristol stool chart (BSC). These criteria will be assessed via the inclusion questionnaire and will be evaluated by the medical supervisor.
* Male and female adults, aged 18-70 years.
* Have a Body Mass Index (BMI) between 18.5 and 30 kg/m2 (self-reported).
* Willing to keep a stable dietary pattern throughout the study.
* Having a smartphone to fill out the daily questionnaires

Exclusion Criteria:

* Having a disease that may interfere with the outcomes of this study, such as a known autonomic disorder, inflammatory bowel disease, coeliac disease, cancer, dialysis patients, chronic kidney failure, depression or hypothyroidism.
* History of intestinal surgery (excluding appendectomy or cholecystectomy) or endometriosis.
* Use of medication that can interfere with the study outcomes, including antidepressants (allowed when it is not subscribed for mental depression), codeine, and antibiotics, as judged by the medical supervisor MD Ben Witteman.
* Use of prescribed laxatives. Over-the-counter laxatives are allowed, but intake should be either stopped before the start of the study or kept stable during the complete study period.
* Use of prebiotics and/or probiotics (should be stopped 4 weeks before the start of the study) and infrequent use of other (fiber) supplements dedicated to bowel function improvements. Some supplements are allowed, but intake should be kept stable during the whole study period (Supplements will be judged by the medical supervisor MD Ben Witteman).
* If applicable: currently pregnant or breastfeeding, or intending to become pregnant during the study, as this can affect stool pattern and wellbeing.
* Participation in another clinical trial at the same time.
* Student or employee working at Food, Health and Consumer Research from Food and Biobased Research, or Department of Human Nutrition & Health, Wageningen University.
* Alcohol intake ≥ 2 (women) or ≥ 4 (men) glasses of alcoholic beverages per day.
* Abuse of illicit drugs, soft drugs, and nitrous oxide.
* Smoking.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Stool frequency | Change after the intervention, measured at week 1, week 4 and week 8
  Number of stools per day will be questioned
Stool consistency | Change after the intervention, measured at week 1, week 4 and week 8
  Will be assessed using the Bristol stool Chart
stool volume | Change after the intervention, measured at week 4 and week 8
  Participants will weigh every stool that they have during 5 days

SECONDARY OUTCOMES:
Constipation severity | during week 1, week 4 and week 8 of the study
  Will be measured using the validated questionnaire PAC-SYM
Irritable Bowel Syndrome severity | during week 1, week 4 and week 8 of the study
  Will be measured using the validated questionnaire IBS-SSS
Constipation related quality of life | during week 1, week 4 and week 8 of the study
  will be measured using the validated questionnaire PAC-QOL
Dietary intake | during week 1, week 4 and week 8 of the study
  will be measured using a validated food frequency questionnaire
Mental wellbeing | during week 1, week 4 and week 8 of the study
  Will be measured using the validated HADS questionnaire
gastro-intestinal complaints | daily for 8 weeks
  will be measured on a visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] JanssenDuijghuijsen L, van den Belt M, Rijnaarts I, Vos P, Guillemet D, Witteman B, de Wit N. Acacia fiber or probiotic supplements to relieve gastrointestinal complaints in patients with constipation-predominant IBS: a 4-week randomized double-blinded placebo-controlled intervention trial. Eur J Nutr. 2024 Aug;63(5):1983-1994. doi: 10.1007/s00394-024-03398-8. Epub 2024 Apr 23. PMID 38653808